CLINICAL TRIAL: NCT06807008
Title: A Novel Pathway to Detect Muscle-invasive Bladder Cancer Based on Integrated Clinical Features and VI-RADS Score on MRI: Results of a Prospective Multicenter Study
Brief Title: A Novel Pathway to Detect Muscle-invasive Bladder Cancer Based on Integrated Clinical Features and VI-RADS Score on MRI
Acronym: VI-RADS
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: VI-RADS
Record Dates: First submitted 2025-01-10; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-12

CONDITIONS: Muscle Invasive Bladder Cancer
Keywords: Magnetic resonance imaging; VI-RADS; Muscle-invasive bladder cancer; Hematuria; Pathway
MeSH Terms: conditions — Hematuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study investigates the clinical, pathological, and radiological features, including the Vesical Imaging-Reporting and Data System (VI-RADS) score, that correlate with muscle-invasive bladder cancer (MIBC). It found that VI-RADS scores, along with other factors, were independent predictors of muscle invasiveness.

DETAILED DESCRIPTION:
The purpose of this study was to determine the clinical, pathological, and radiological features, including the Vesical Imaging-Reporting and Data System (VI-RADS) score, independently correlating with muscle-invasive bladder cancer (BCa), in a multicentric national setting. Patients with BCa suspicion were offered magnetic resonance imaging (MRI) before trans-urethral resection of bladder tumor (TURBT). According to VI-RADS, a cutoff of ≥ 3 or ≥ 4 was assumed to define muscle-invasive bladder cancer (MIBC). Trans-urethral resection of the tumor (TURBT) and/or cystectomy reports will be compared with preoperative VI-RADS scores to assess accuracy of MRI for discriminating between non-muscle-invasive versus MIBC. Performance will be assessed by ROC curve analysis. Two univariable and multivariable logistic regression models were implemented including clinical, pathological, radiological data, and VI-RADS categories to determine the variables with an independent effect on MIBC.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of bladder tumor,
* positive urinary cytology,
* suspected bladder neoplasm identifed by ultrasound of the urinary tract and/or cystoscopy and/or CT scan of the abdomen-pelvis.

Exclusion Criteria:

* history of prior urinary tract neoplasms,
* impossibility of achieving appropriate bladder distension,
* concomitant diagnosis of carcinoma in situ (CIS),
* no detectable lesion on MRI
* any contraindication to MRI (low renal function, MR unsafe medical devices etc.)
* any contraindication to spinal and general anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter prospective observational study received formal approval from the Institutional Review Board and Ethics Committee of each participating center. All patients were informed of the experimental nature of this study and gave written informed consent. All patients with suspected BCa were referred to four different centers (Sapienza University of Rome [center #1], Istituto Nazionale Tumori "Regina Elena" in Rome [center #2], Azienda Ospedaliera Universitaria Santa Maria della Misericordia in Udine [center #3], and Azienda Ospedaliera Universitaria in Bologna [center #4]), between January 2020 and May 2021, and underwent bladder MRI.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
The accuracy of the VI-RADS (Vesical Imaging-Reporting and Data System) score in predicting muscle-invasive bladder cancer (MIBC) preoperatively using MRI. | 6 weeks
  In order to evaluate the diagnostic accuracy of the VI-RADS score in correctly differentiating non-muscle from muscle-invasive bladder disease at first diagnosis, diagnostic performance variables (sensitivity, specificity, accuracy, positive and negative predictive value, area under the curve, and ROC curves) will be calculated both overall over all participating centers and independently for different centers.
  The gold standard for differential diagnosis between NMIBC and MIBC will be represented by:
  * TURBT in those cases then classified as low-risk NMIBC;
  * Re-TURBT in those patients who are candidates for Re-TURBT according to the guidance provided by the EAU guidelines [14-15];
  * TURBT and/or radical cystectomy in those cases classified as MIBC (≥T2).

SECONDARY OUTCOMES:
The correlation between specific clinical features and MIBC. | 6 weeks
  The correlation between specific clinical features (e.g., lesion size, presence of hydronephrosis) and MIBC. These factors were evaluated in conjunction with VI-RADS scores to refine diagnostic and predictive models

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Schiavina, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (4):
- Italy (4):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - AOU Policlinico Umberto I - Sapienza University of Rome, Roma, Italy
  - Regina Elena" National Cancer Institute, Roma, Italy
  - Santa Maria della Misericordia University Hospital in Udine, Udine, Italy

IPD SHARING:
Plan to Share IPD: No